CLINICAL TRIAL: NCT06873256
Title: Evaluation of the Hospital Pathway for Frail Elderly Patients Hospitalised for Pathologies Leading to Medical Decompensation
Acronym: FRAGIL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-CHITS-011
Record Dates: First submitted 2025-02-21; First posted 2025-03-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Frail Elderly People Hospitalized
Keywords: Elderly person; Weakness; Addressing; Nursing home; 911
MeSH Terms: conditions — Asthenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Frail patients hospitalized for medical decompensation

SUMMARY:
People aged over 75 account for 25% of emergency department visits in the Provence Alpes Côte d'Azur region. Depending on the facility, around 50% of these patients are discharged home without being hospitalised. Yet the scientific literature highlights the frequent deterioration in the physical and mental state of the elderly during a visit to the emergency department: discomfort on the stretcher, waiting, loneliness and disorientation are the causes, and therefore increase co-morbidity. Very few studies have been carried out to date to compare the impact on frailty risk factors of direct admission to hospital versus admission via emergency service for a frail elderly population. Studies are usually based on a population aged over 75 as the sole criterion, which no longer corresponds to the definition of a frail elderly person. What's more, there are major challenges in coordinating hospital and outpatient care to optimise resources.

The aim is to assess whether the creation of new care pathways, requiring considerable human and financial resources, will improve the care of frail elderly people. In order to assess the benefits of the systems set up at the hospital this study will compare the outcome of frail elderly people (≥ 75 years old with a geriatric score ≥ 8) hospitalised for medical decompensation pathologies according to their mode of admission, the management of their dependency and their accessibility to the attending physician, whether in individual accommodation or in an Residential Establishment for Dependent Elderly People.

This is a regional multicentre, observational, prospective and retrospective study looking at the future of frail elderly people hospitalised at the hospital during 2024/2025 (from 01/09/2024 to 01/03/2025).

The study will be conducted retrospectively, including patients hospitalised since 1st September 2024, and prospectively, including patients over time until the end of the inclusion period (01/03/2025). Patients will be followed for 90 days after hospitalisation, i.e. data will be collected until 01/06/2025.

Justification of the public interest

This research could make it possible to identify new protective factors against deterioration in the frail elderly, other than direct admission to a hospital ward, which would require fewer human and material resources, such as an Mobile Geriatric Team or a stay in a Short-Term Hospitalization Unit.

If direct admissions lead to fewer patients being admitted back to hospital, this could encourage existing medical and surgical specialties outside geriatrics and support geriatric assessment.

Lastly, this research would make it possible to draw up an inventory of the frailty of the elderly in the Toulon conurbation, in order to optimise the screening of frail elderly people in conjunction with the territorial care coordination west var region.

Data collection begins as soon as the frail elderly person is hospitalised and continues for up to 90 days after the start of hospitalisation (retrospectively and prospectively).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 75 years;
* Patient cared for at the Intercommunal Hospital Center of Toulon-La Seyne sur Mer (Sainte Musse and Georges Sand hospitals) between 01/09/2024 and 01/03/2025 and presenting a geriatric score ≥ 8 (score defined by multidisciplinary work);
* Patient requiring hospitalisation for medical decompensation.

Exclusion Criteria:

* Patient with acute pathologies requiring admission to the intensive care unit;
* Patient whose care is in the field of traumatology in isolation;
* Patient's refusal to take part in the research.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Frail elderly people hospitalized
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
The main objective was to assess the 90-day morbidity and mortality of frail elderly people hospitalized, depending on their mode of hospitalization. | 3 months
  The primary endpoint was early re-hospitalization or death within 90 days, depending on the mode of hospitalization (short-term hospital unit, direct admissions and passage via the emergency department).

SECONDARY OUTCOMES:
To assess the 30-day morbidity and mortality of frail elderly people hospitalized according to their mode of hospitalization. | 1 month
  Number of early re-hospitalization or death within 30 days, depending on the mode of hospitalization (short-term hospital unit, direct admissions and passage via the emergency department).
Evaluate the prognosis of frailty at a distance, based on the presence of a Mobile Geriatric Team during hospitalization and on the implementation of an assistance plan in conjunction with a hospital social worker, enabling a safe return home. | 1 month
  Number of early re-hospitalizations or deaths at 30 days, depending on the presence of a Mobile Geriatric Team during hospitalization (Yes/No) and the request to set up/organize an assistance plan in conjunction with a social worker (Yes/No/Not applicable).
Evaluate the prognosis of frailty at a distance, based on the presence of a Mobile Geriatric Team during hospitalization and on the implementation of an assistance plan in conjunction with a hospital social worker, enabling a safe return home. | 3 months
  Number of early re-hospitalizations or deaths at 90 days, depending on the presence of a Mobile Geriatric Team during hospitalization (Yes/No) and the request to set up/organize an assistance plan in conjunction with a social worker (Yes/No/Not applicable).
For the sub-group of patients referred from nursing homes, assess the time between the last General Practitioner referral and hospitalization. | 1 year before hospitalization
  Time in days between last medical contact with a general practitioner and hospitalization. The date of the last medical contact will be retrieved from the Residential establishment for dependent elderly people's Emergency Liaison File
Evaluate the proportion of frail patients who have been specifically identified by the territorial care coordination teams prior to hospitalization. | 1 year before hospitalization
  Rate of frail patients identified by the territorial care coordination West Var region (following a report made by a nurse, a doctor or a care assistant) prior to hospitalization, compared to the rate of frail patients hospitalized.
Analyze the patient's destination at the end of the initial hospitalization | Up to 1 month
  The following destinations at discharge from hospitalization will be analyzed: Follow-up and rehabilitation care / Residential establishment for dependent elderly people / Home / Death during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marc FOURNIER, MD, Study Director — Centre Hospitalier Intercommunal Toulon- La Seyne sur mer
Locations (1):
- Centre Hospitalier Intercommunal Toulon-La Seyne sur Mer, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The predictive validity of frailty status for hospitalization and mortality. In: The predictive validity of the state of frailty for hospitalization and mortality. Toulouse: The 2016 Gerontological Year; 2016. p. 49 49.Brun M. C3S Coordination Support Sc — https://dumas.ccsd.cnrs.fr/dumas-03643709
- See also: Report of the Hospital and Elderly Persons Workshop — https://sante.gouv.fr/IMG/pdf/synthese_atelier_10_hopital_et_personne_agee_14_fev_2018_3_.docx.pdf
- See also: ICOPE - A program to prevent addiction [Internet]. 2023 [cited 2024 Sep 22]. — https://sante.gouv.fr/IMG/pdf/icope_cahier_des_charges_220322.pdf
- See also: Elderly people in the emergency room: a more fragile health requiring longer care: Studies and results 2017; N°1008 Electronic ISSN 1146-9129. — https://www.drees.solidarites-sante.gouv.fr/publications/etudes-et-resultats/les-personnes-agees-aux-urgences-une-sante-plus-fragile
- See also: Hospital emergencies in 2023: what organizations for patient care? Studies and results 2024 N°1305; Electronic ISSN 1146-9129. — https://www.drees.solidarites-sante.gouv.fr/publications-communique-de-presse/etudes-et-resultats/240711_ER_UrgencesHospitalieres2023